CLINICAL TRIAL: NCT04095962
Title: Body and Brain: Effects of a Multicomponent Exercise Intervention on Physical and Cognitive Function of Older Adults With Dementia
Brief Title: Effects of a Multicomponent Exercise Intervention on Physical and Cognitive Function of Older Adults With Dementia
Acronym: Body&Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BB01
Record Dates: First submitted 2019-08-20; First posted 2019-09-19 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-09

CONDITIONS: Dementia; Alzheimer Disease; Vascular Dementia; Neurocognitive Disorders
Keywords: Functionality; Multimodal; Cognition
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular; Neurocognitive Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Training protocol will be held for 6 months, twice per week/ 60 min per sessions.
  Interventions: Other: Exercise
- Control Group (No Intervention): Participants in the control group will receive monthly sessions regarding physical activity and health related topics as a complement to standard care. No specific exercise intervention will be conducted for this group.

INTERVENTIONS:
Other: Exercise — The MT program will be conducted for 6 months, twice a week in 60 minutes sessions. Sessions will be divided in warm-up (10 minutes, including slow walk, postural and mobility exercises for general activation, and stretching exercises), specific training (35-45 minutes, including balance/coordination training, strength and aerobic exercises) and cool down (5 minutes with breathing and stretching exercises for the main worked joints and muscles) following the main guidelines recommended by the American College of Sports Medicine [18] and the WHO [19].
  Other Names: Multicomponent training
  Arms: Experimental Group

SUMMARY:
Dementia is a leading cause of death and disability that was declared as one of the greatest health and social care challenges of the 21st century. Regular physical activity and exercise have been proposed as a non-pharmacological strategy in disease prevention and management. Multicomponent Training (MT) combines aerobic, strength, balance, and postural exercises and might be an effective training to improve both functional capacity and cognitive function in individuals with dementia (IwD). Nevertheless, data on the effects of MT in IwD are still limited and the extent to which IwD can retain improvements after an exercise intervention still needs to be elucidated. The aim of "Body & Brain" study is to investigate the effects of a 6-month MT intervention and 3-month detraining on the physical and cognitive function of IwD. Additionally, we aim to explore the impact of this intervention on psychosocial factors and physiologic markers related to dementia.

DETAILED DESCRIPTION:
Although exercise interventions for IwD seem to be feasible and well tolerated, resulting in positive effects on ADL functionality for people at mild-to-moderate stages [1, 2], the therapeutic role of physical activity, particularly exercise, after dementia diagnosis still needs further evidence [3-5], - especially when considering community-based contexts and caregivers as participants on exercise sessions [6]. It also matters to highlight that the dose-dependent relationship remains unclear [1, 7, 8]. Therefore, research is needed to identify the triad: stage/type of dementia, FITT variables (frequency, intensity, type, and time) of exercise intervention, and target outcome [7, 9]. Regarding exercise modality, Multicomponent Training (MT) [10] - combining aerobics, strength and balance exercises - seems to be effective at improving functional and cognitive performances in older adults with neurodegenerative disorders, particularly dementia [11-13]. Exercise programs previously developed by our group confirmed that a 6-month MT intervention can positively impact the physical and cognitive function of institutionalized older adults with AD [14, 15] and can be beneficial in physical fitness and ADL functionality performance among community-dwelling patients [9, 16]. However, the extent to which IwD can retain these improvements after the cessation of MT intervention still need to be elucidated [17] in order to understand how detraining affects functionality and cognition following the cessation of MT stimulus.

This study is a quasi-experimental controlled trial using a parallel-group design. The study sample consists of community-dwelling individuals aged ≥ 60 years who are clinically diagnosed with dementia or major neurocognitive disorder. Participants will be either allocated into the intervention group or the control group. The intervention group will participate in MT biweekly exercise sessions, whereas the control group will receive monthly sessions regarding physical activity and health-related topics for 6 months. The main outcomes will be physical function as measured by the Short Physical Performance Battery (SPPB) and cognitive function evaluated using the Alzheimer Disease Assessment Scale - Cognitive (ADAS-Cog) at baseline, after 6-months and 3-months after the end of intervention. Secondary outcomes will be body composition, physical fitness, daily functionality, quality of life, neuropsychiatric symptoms and caregiver's burden. Cardiovascular, inflammatory and neurotrophic blood-based biomarkers, and arterial stiffness will also be evaluated in subsamples.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged ≥ 60 years capable of walking autonomously without an assistive device or human assistance;
* Individuals diagnosed with dementia or major neurocognitive disorder using accepted diagnostic criteria such as that established by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR or DSM-5), ICD-10, or the NINCDS-ADRDA; by a physician for at least for 6-months.

Exclusion Criteria:

* Individuals diagnosed with certain disorders or conditions in which exercise is contraindicated such as unstable or ongoing cardiovascular and/or respiratory disorder;
* Hospitalized individuals and/or recovering from surgery or rehabilitation;
* Individuals presenting an advanced stage of dementia (e.g., scored 3-points in CDR or ≤ 10 points on MMSE) that could affect physical performance in the exercise training sessions or testing procedures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on Short Physical Performance Battery (SPBB) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The Short Physical Performance Battery (SPPB) is a standardised assessment tool of lower limb function, testing 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4, total score from 0 (poor performance) to 12 (best performance).
Change from Baseline on Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  To evaluate cognitive function with a total scoring ranging between 0 - 68. A score of 68 represents the most severe impairment and 0 represents the least impairment.

SECONDARY OUTCOMES:
Change from Baseline on 30-second Chair-stand Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical fitness is going to be measured via the Senior Fitness Test (SFT).This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively), aerobic endurance (2-minute step test), and agility/dynamic balance (8-foot up-and-go test).
  Lower body strength was measured using the 30 s chair stand test. Participants were asked to sit in a 43-cm armless chair with their arms crossed at the wrists and held against the chest. The score was the total number of stands executed correctly within 30 s.
Change from Baseline on 30-second Arm Curl Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical fitness is going to be measured via the Senior Fitness Test (SFT).This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively), aerobic endurance (2-minute step test), and agility/dynamic balance (8-foot up-and-go test).
  Upper body strength was assessed using the arm curl test. Participants performed as many biceps curls as possible in 30 s, using a dumbbell (3.63 kg and 2.27 kg for men and women, respectively). The score was the total number of hand-weight curls performed through the full range of motion within 30 s.
Change from Baseline on 2-minute Step Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical fitness is going to be measured via the Senior Fitness Test (SFT).This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively), aerobic endurance (2-minute step test), and agility/dynamic balance (8-foot up-and-go test).
  Cardiorespiratory fitness was measured using 2-min step test. Participants were asked to raise each knee to a point midway between the patella (kneecap) and iliac crest (top hip bone). The score was the number of times the right knee reaches the required height.
Change from Baseline on 8-Foot Up and Go Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical fitness is going to be measured via the Senior Fitness Test (SFT).This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively), aerobic endurance (2-minute step test), and agility/dynamic balance (8-foot up-and-go test).
  Participants were asked to as quickly as possible, in a sitting position, stand up, walk 8-foot distance (2,44 meters), turn the cone marker around and return to the seated position. The time, in seconds, necessary to complete this test was registered.
Change from Baseline on Back Scratch Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical fitness is going to be measured via the Senior Fitness Test (SFT).This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively), aerobic endurance (2-minute step test), and agility/dynamic balance (8-foot up-and-go test).
  Upper-body flexibility was measured through the back-scratch test. The participants were asked to, in standing position, place the preferred hand over the same shoulder, reaching down the middle of the back as far as possible - elbow pointed up. Then, the participants were asked to place the other arm around the back of the waist with the palm up and in attempt to touch (or overlap) the extended middle fingers of both hands. The nearest distance (in centimeters) was measured between the tips of the middle fingers (minus or plus, depending if overlapping or not)
Change from Baseline on Sit and reach Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical fitness is going to be measured via the Senior Fitness Test (SFT).This physical battery includes lower and upper-body strength (30-second chair stand and 30-second arm curl tests, respectively), lower and upper-body flexibility (chair sit-and-reach and back scratch tests, respectively), aerobic endurance (2-minute step test), and agility/dynamic balance (8-foot up-and-go test).
  The chair sit-and-reach test was used to assess lower-body flexibility. Participants were asked to sit at the front edge of a chair and with one leg extended (dominant) reach the toward toes as far as possible, bending the upper body forward at the hip joint. The other leg must be bent and slightly off to one side with the foot flat on the floor. The number of centimeters (plus or minus) were registered between the extended fingers (hands overlapping) and the tip of the toe - maintaining the position for at least 2 seconds.
Change from Baseline on Modified Bruce Treadmill Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  This sub-maximal test with incremental protocol including seven stages and performed on a treadmill. To assess Peak oxygen uptake (VO2 peak), standard an open-circuit spirometer technique (Cosmed K4b2, Cosmed, Rome, Italy) will be used.
Change from Baseline on One Leg Balance Test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The static balance will be measured with the One Leg Balance Test. Participants will be asked to choose a leg to stand on, flex the opposite knee and balance on one leg as long as possible. The time (in seconds) standing unsupported will be recorded.
Change from Baseline on Handgrip test | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Handgrip strength will be obtained with a Jamar Plus + Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA).Measurements will be carried out following the American Society of Hand Therapists recommendations, and each participant will perform three attempts with a pause of 1 min between them. The maximum value, in kilograms of force (kgf), of the three measurements with the dominant hand will be registered.
Change from Baseline on Appendicular Skeletal Muscle Mass Index (ASMI) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Appendicular Skeletal Muscle Mass Index (ASMI), which is the sum of muscle masses of the four limbs described as appendicular skeletal muscle mass adjusted for height (kg/m2), will be analyzed with Dual Energy X-ray Absorptiometry (DXA) (Hologic QDR 4500, Explorer model, version 12.4).
Change from Baseline on Body mass, fat-free mass, fat mass | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Body mass (kg), fat-free mass (kg) and fact mass (kg) will be analyzed with Dual Energy X-ray Absorptiometry (DXA) (Hologic QDR 4500, Explorer model, version 12.4)
Change from Baseline on Barthel Index (BI) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  To evaluate independence on performing basic activities of daily living, ranging from 0-100 and with higher scores representing increased functionality.
Change from Baseline on Lawton & Brody (IADL) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Assessment of instrumental activities of daily life. It evaluates the following categories and subcategories: A. Ability to Use Telephone; B. Shopping; C.Food Preparation; D.Housekeeping; E. Laundry; F. Mode of Transportation; G. Responsibility for Own Medications; H. Ability to Handle Finances. Range 0-8. Lower scores are indicative of increased difficulties to independently perform instrumental activities.
Change from Baseline on Mini-Mental State Examination (MMSE) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The Mini Mental State Examination (MMSE) a widely used test of cognitive function among older adults will be used and consists of a 30-item instrument (with higher scores indicating better cognitive performance) that is organized in six cognitive domains - orientation, retention, attention and calculation, delayed recall, language, and visuo-constructive ability.
Change from Baseline on Trail-making test (TMT) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The executive functions will be assessed with the Trail Making Test part A - attention, visual scanning, speed of eye-hand coordination, and information processing; and part B - working memory and the ability to switch between different stimuli. Time and number of errors will be registered.
Change from Baseline on Neuropsychiatric inventory (NPI) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  NPI is used to determine the frequency and severity of behavioral and psychological symptoms of dementia (BPSD) with a total score ranging from zero to 144 points with high scores corresponding to worsening of BPSD.
Change from Baseline on Quality of Life in Alzheimer's Disease scale (QoL-AD) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The QoL-AD will be used to measure the dementia participants' quality of life. The questionnaire includes 13 items such as physical health, energy, mood, memory, family, marriage, friends, and ability to do things for fun. The QoL-AD provides the participant and the caregiver reports of the participant's QoL and is scored on a 4-point Likert-type scale ranging from 1 to 4 (excellent), with total scores ranging between 13 and 52 point, and higher scores indicating better quality of life.
Change from Baseline on Caregiver subjective burden (CarerQol-7D) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The Care-related Quality of Life instrument (CarerQol) will be used to address subjective burden (CarerQol-7D). The subjective burden is measured in seven dimensions: fulfillment, relational problems, mental health, daily activities problems, physical health and support. Total CarerQol-7D score ranges from 0 to 14 points with higher scores indicating better caregiving situation.
Caregiver subjective well-being (CarerQol-VAS) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  The Care-related Quality of Life instrument (CarerQol) will be used to address caregivers' well-being (CarerQol-VAS), using a visual analogue scale to ask about happiness between 0 (completely unhappy) and 10 (completely happy).
Change from Baseline on Blood triglycerides (TG), total cholesterol (TC), Low-density lipoprotein cholesterol (LDL-C) and high-density lipoprotein cholesterol (HDL-C) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Determination of TG (mg/dL), TC (mg/dL),LDL-C (mg/dL), HDL-C (mg/dL) concentrations in plasma.
Change from Baseline on Circulating levels of Glycated Hemoglobin (HbA1c) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Determination of HbA1c(μg/mL) concentrations in blood.
Change from Baseline on Circulating levels of Interleukin-6 (IL-6),Interleukin-8 (IL-8), Interleukin-10 (IL-10) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Plasma IL-6 (pg/ml), IL-8 (pg/ml), IL-10 (pg/ml) concentrations will be measured using V-PLEX Human Biomarker 40-Plex Kit pro-inflammatory.
Change from Baseline on Circulating levels of C-Reactive Protein (CRP) and Tumor Necrosis Factor (TNF-alfa) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Plasma CRP (μg/mL) and TNF-alfa (μg/mL) concentrations will be measured using V-PLEX Human Biomarker 40-Plex Kit pro-inflammatory.
Change from Baseline on Circulating levels of free brain-derived neurotrophic factor (BDNF),Vascular Endothelial Growth Factor (VEGF), intercellular adhesion molecule 1 (sICAM-1), vascular cell adhesion molecule-1 (sVCAM-1), metalloproteinase-9 (MMP-9) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  BDNF (pg/ml), VEGF (pg/ml), sICAM-1 (pg/ml), sVCAM-1 (pg/ml), MMP-9 (pg/ml) concentrations will be analysed using the ELISA method (enzyme-linked immunosorbent assay).
Change from Baseline on Circulating levels of Insulin-like growth factor-1 (IGF-1) | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Plasma IGF-1 (ng/ml) concentrations will be measured by the DiaSorin using a LIAISON ® kit and analysed by CLIA method.
Change from Baseline on Systolic and Diastolic Blood Pressure | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Systolic and Diastolic Blood Pressure (mmHg) will be measured using a digital sphygmomanometer.
Change from Baseline on Arterial stiffness | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Arterial stiffness is going to be measured as carotid-femoral pulse wave velocity (cfPWV) using applanation tonometry (SphygmoCor, AtCor Medical, Australia). Procedures will follow international guidelines. In brief, sequential and consecutive carotid and femoral pressure waves are going to be registered together with the electrocardiogram, which will serve as a reference to calculate the transit time between the recording's sites. The distance traveled by the pressure wave will be the direct distance between the recording points at the femoral and carotid arteries, corrected by the factor 0.8. The value of cfPWV is going to be calculated as the direct distance (in meters) divided by the transit time (in seconds). All measurements will be performed in duplicate by the same trained researcher.

OTHER OUTCOMES:
Change from Baseline on Daily Physical Activity levels | Assessment at baseline, immediately after 6 months of intervention, and at 3 months follow-up for experimental and control groups
  Physical activity levels will be collected with the activity monitors GT3X+ (ActiGraph), located at the waist, to measure the activity intensity (counts per minute) during one week.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Carvalho, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Sports of University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques-Aleixo I, Sampaio A, Bohn L, Machado F, Barros D, Ribeiro O, Carvalho J, Magalhaes J. Neuropsychiatric Symptoms are Related to Blood-biomarkers in Major Neurocognitive Disorders. Curr Aging Sci. 2024;17(1):74-84. doi: 10.2174/1874609816666230816090934. PMID 37904566
- [Derived] Borges-Machado F, Teixeira L, Carvalho J, Ribeiro O. Does Multicomponent Physical Exercise Training Work for Dementia? Exploring the Effects on Cognition, Neuropsychiatric Symptoms, and Quality of Life. J Geriatr Psychiatry Neurol. 2023 Sep;36(5):376-385. doi: 10.1177/08919887221149152. Epub 2022 Dec 27. PMID 36574616
- [Derived] Borges-Machado F, Barros D, Teixeira L, Ribeiro O, Carvalho J. Contribution of a multicomponent intervention on functional capacity and independence on activities of daily living in individuals with neurocognitive disorder. BMC Geriatr. 2021 Nov 3;21(1):625. doi: 10.1186/s12877-021-02591-2. PMID 34732148
- [Derived] Borges-Machado F, Barros D, Teixeira L, Ribeiro O, Carvalho J. Health-related physical indicators and self-rated quality of life in older adults with neurocognitive disorder. Qual Life Res. 2021 Aug;30(8):2255-2264. doi: 10.1007/s11136-021-02828-y. Epub 2021 Mar 28. PMID 33778911
- [Derived] Carvalho J, Borges-Machado F, Barros D, Sampaio A, Marques-Aleixo I, Bohn L, Pizarro A, Teixeira L, Magalhaes J, Ribeiro O. "Body & Brain": effects of a multicomponent exercise intervention on physical and cognitive function of adults with dementia - study protocol for a quasi-experimental controlled trial. BMC Geriatr. 2021 Mar 4;21(1):156. doi: 10.1186/s12877-021-02104-1. PMID 33663414
- [Derived] Sampaio A, Marques-Aleixo I, Seabra A, Mota J, Carvalho J. Physical exercise for individuals with dementia: potential benefits perceived by formal caregivers. BMC Geriatr. 2021 Jan 6;21(1):6. doi: 10.1186/s12877-020-01938-5. PMID 33407194